CLINICAL TRIAL: NCT06502678
Title: Systemic Sclerosis: the Role of Autoantibodies and Their Blockade in the Disease Pathogenesis. In Vitro and in Vivo Experimental Models
Brief Title: AUTOANTIBODIES AND SYSTEMIC SCLEROSIS
Acronym: AUTO
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Marco Matucci-Cerinic, MD PhD, IRCCS Ospedale San Raffaele
Other Study IDs: AUTO
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Understand Pathogenicity of SSc-specific Antibodies in SSc and the Effect of Antibody Blockade in Vitro

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Fcr blocker of autoantibodies — in vitro assays, combined with multi-omics approach and in vitro experimental models, will gain insights into the pathogenesis of Systemic Sclerosis (SSc)dissecting the consequences of treatment with Fcblocker on functional and phenotypic cell behavior. Healthy microvascular endothelial cells, fibroblasts and monocytes will be challenged with serum and autoantibodies prior to or upon treatment with Efgartigimod in order to assess both the prevention and the recovery capacity of the FcR blocker. The putative modulatory effect of Efgartigimod on vascular remodeling, endothelial-to-mesenchymal transition, fibroblast-to-myofibroblasts transition and monocyte behavior will be evaluated in in-vitro consolidated assays. Integrated Omics analyses will support and complement the in vitro findings by unveiling potential prognostic signatures and by identifying specific treatment-related profiles that might guide the modulation of the drug usage in order to maximize its beneficial effect

SUMMARY:
Established in vitro assays, combined with state-of-the-art multi-omics approaches and innovative in vitro experimental models, will gain insights into the mechanistic bases underlying Systemic Sclerosis (SS) pathogenesis and will dissect the consequences of treatment with Efgartigimod on functional and phenotypic cell behaviors. Healthy microvascular endothelial cells, fibroblasts and monocytes will be challenged with serum and autoantibodies prior to or upon treatment with Efgartigimod in order to assess both the prevention and the recovery capacity of the FcR blocker. The putative modulatory effect of Efgartigimod on vascular remodeling, endothelial-to-mesenchymal transition, fibroblast-to-myofibroblasts transition and monocyte behavior will be evaluated in in-vitro consolidated assays. Integrated Omics analyses will support and complement the in vitro findings by unveiling potential prognostic signatures and by identifying specific treatment-related profiles that might guide the modulation of the drug usage in order to maximize its beneficial effects.

ELIGIBILITY:
Inclusion Criteria:

* positivity of autoantibodies

Exclusion Criteria:

* pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: systemic sclerosis patients characterised by the autoantibody positivity
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Verify if Fcblocker can block the pathogenic activity of autoantibodies | 24 months
  To assess both the prevention and the recovery capacity of the FcR blocker in different kind of cells submitted to the specific autoantibody. microvascular endothelial cells and fibroblasts

IPD SHARING:
Plan to Share IPD: No